CLINICAL TRIAL: NCT02988128
Title: NeuroVascular Product Surveillance Registry (PSR) Platform
Brief Title: Neurovascular Product Surveillance Registry
Acronym: INSPIRE
Status: Recruiting | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Collaborators: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT16056/17077/24028/22032
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Intracranial Aneurysm; Stroke, Ischemic
Keywords: Embolization Device; Flow Diverter; Intrasaccular device; Vascular Reconstruction Device; Ruptured Intracranial Aneurysm; Unruptured Intracranial Aneurysm; Large Vessel Occlusion; Stent Retriever; Aspiration Catheter; Revascularization Device
MeSH Terms: conditions — Intracranial Aneurysm; Ischemic Stroke | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Intracranial aneurysm: Patients undergoing treatment for intracranial aneurysms (IA) with Medtronic market approved device(s).
  Interventions: Device: Treatment for intracranial aneurysms
- Acute Ischemic Stroke: Patients undergoing treatment for acute ischemic stroke (AIS) with Medtronic market approved device(s).
  Interventions: Device: Treatment for Acute Ischemic Stroke

INTERVENTIONS:
Device: Treatment for intracranial aneurysms — Embolization of aneurysms
  Groups: Intracranial aneurysm
Device: Treatment for Acute Ischemic Stroke — Revascularization of an intracranial blood vessel
  Groups: Acute Ischemic Stroke

SUMMARY:
Post market surveillance registry

DETAILED DESCRIPTION:
An observational, prospective, multi-center, single-arm registry to provide continuing evaluation and periodic reporting of safety and effectiveness of Medtronic Neurovascular market-released products used in the treatment of Intracranial aneurysms and Acute Ischemic Stroke.

MDT16056 and MDT17077 are conducted under the Product Surveillance Registry (NCT01524276).

ELIGIBILITY:
For MDT16056 and MDT17077

Inclusion Criteria:

* Patient or legally authorized representative (LAR) provides authorization and/or consent per institution and geographical requirements
* Patient has, or is intended to receive or be treated with, an eligible Medtronic product
* Patient is consented within the enrollment window of the therapy received, as applicable
* Patient is at least 18 years of age at time of enrollment.

Exclusion Criteria:

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results
* Female patient who is known to be pregnant or is breastfeeding or wishes to become pregnant during participation in the study.

For MDT24028 and MDT22032:

General Inclusion Criteria:

* Patient or legally authorized representative (LAR) provides authorization and/or consent per institution and geographical requirements.
* Patient is treated or intended to be treated with an eligible Medtronic Neurovascular product.
* Patient is an adult per local law at time of consent. Medtronic Business Restricted This document is electronically controlled CONFIDENTIAL 056-F275 Rev F Clinical Investigation Plan Template

General Exclusion Criteria:

* Patient who may be unable to complete the study follow-up
* Patient with any contraindications per the applicable Instructions for Use document
* Female patient who is known to be pregnant or is breastfeeding or wishes to become pregnant during participation in the study
* Patient is currently enrolled in, or plans to enroll in, any concurrent drug/device study that may confound the study results.

Additional criteria may be required, refer to cohort-specific Addendum, as applicable, for further guidance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intracranial aneurysms: Patients requiring treatment for intracranial aneurysms with Medtronic market-approved flow diverters, intrasaccular devices, vascular reconstruction devices and/or ancillary devices are eligible for the registry.
  Acute Ischemic Stroke: Patients requiring treatment with Medtronic market approved stent retrievers and/or aspiration devices, and/or ancillary devices for the treatment of acute ischemic stroke due to intracranial vessel occlusion are eligible for enrollment in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2032-08 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
The clinical success rate defined as complete occlusion of target aneurysm without retreatment or significant artery stenosis (≤ 50%). | 1 year
  For Intracranial Aneurysm the primary outcome is the clinical success rate defined as complete occlusion of target aneurysm without retreatment or significant artery stenosis (≤ 50%).
Functional Independence: mRS score ≤ 2 | 90 days
  For Acute ischemic stroke the primary outcome is functional Independence: modified Rankin Scale (mRS) score ≤ 2

CONTACTS AND LOCATIONS:
Overall Officials: Markus Holtmannspotter, MD, Study Chair — Klinikum Nürnberg Süd; Laurent Spelle, MD, Study Chair — Hôpital Bicêtre, Service de Neuroradiologie Interventionnelle Adulte et Pédiatrique; Jens Fiehler, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf; István Szikora, MD, Study Chair — National Institute of Clinical Neurosciences; Mario Galdamez, MD, Study Chair — Hospital Clínico Universitario de Valladolid; Saleh Lamin, MD, Study Chair — Queen Elisabeth Hospital, Neuroradiology; Francis Turjman, MD, Study Chair — Hôpital Pierre Wertheimer; Christophe Cognard, MD, Study Chair — CHU Toulouse - Hôpital Purpan; Markus Möhlenbruch, MD, Study Chair — University Hospital Heidelberg; Marc Ribó, MD, Study Chair — Hospital Vall d'Hebron; Pasquale Mordasini, MD, Study Chair — Inselspital - Universitätsspital Bern; Sanjeev Nayak, MD, Study Chair — University Hospitals of North Midlands NHS Trust - Royal Stoke University Hospital; Riitta Rautio, MD, Study Chair — Turun Yliopistollinen keskussairaala; Monika Killer-Oberpfalzer, MD, Study Chair — Universitätsklinikum Christian Doppler Klinik Salzburg
Locations (99):
- ENERI, Buenos Aires, Argentina
- Gold Coast University Hospital, Southport, Australia
- Universitätsklinikum Christian Doppler Klinik Salzburg, Salzburg, Austria
- Belgium (2):
  - Ziekenhuis Oost Limburg - Campus Sint-Jan, Genk
  - Universitair Ziekenhuis Gent, Ghent
- China (18):
  - Xuanwu Hospital Capital Medical University, Beijing
  - Chongqing University Three Gorges Hospital, Chongqing
  - First Affiliated Hospital of Jiamusi University, Jiamusi
  - The Affiliated Hospital of Jinggangshan University, Ji’an
  - Kaifeng Central Hospital, Kaifeng
  - Liaocheng People's Hospital, Liaocheng
  - Lishui Municipal Central Hospital, Lishui
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - The Second Nanning Peoples Hospital, Nanning
  - Panzhihua Central Hospital, Panzhihua
  - Qujing First Peoples Hospital, Qujing
  - Yangpu District Central Hospital Shanghai Yangpu Hospital Tongji University, Shanghai
  - Shanxi Cardiovascular Hospital, Taiyuan
  - The First Affiliated Hospital Of Xi'an Jiaotong University, Xi'an
  - The First Peoples Hospital of Xianyang, Xianyang
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou
  - Zhuhai Peoples Hospital, Zhuhai
  - Zhumadian Central Hospital, Zhumadian
- Rigshospitalet, Copenhagen, Denmark
- Turun Yliopistollinen keskussairaala, Turku, Finland
- France (21):
  - CHU Besancon - Hôpital Jean Minjoz, Besançon
  - CHU de Bordeaux - Centre Universitaire Pellegrin, Bordeaux
  - CHU Brest, Hôpital de la Cavale Blanche, Brest
  - Hôpital Pierre Wertheimer, Bron
  - CHU de Caen, Caen
  - Centre Hospitalier Universitaire de Clermont-Ferrand - Gabriel-Montpied, Clermont-Ferrand
  - CHU Dijon Bourgogne, Dijon
  - AP-HP Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU Limoges - Hôpital Dupuytren, Limoges
  - Hôpital de la Timone-CHU de Marseille, Marseille
  - CHU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - CHU de Nancy - Hôpital Central, Nancy
  - CHU de Nantes Hôpital Laennec, Nantes
  - GHU Paris Psychiatrie & Neurosciences, Paris
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Hôpital de la Pitié Salpétrière, Paris
  - CHU Reims Hôpital Maison Blanche, Reims
  - CHU Hôpitaux de Rouen - Hôpital Charles Nicolle, Rouen
  - CHU Toulouse - Hôpital Pierre-Paul Riquet, Toulouse
  - CHRU de Tours - Hôpital Brettoneau, Tours
  - Centre Hospitalier Bretagne Atlantique Vannes - Auray, Vannes
- Germany (11):
  - Klinikum Augsburg, Augsburg
  - Charité Universitätsmedizin Berlin -Campus Charite, Berlin
  - Knappschaftskrankenhaus Bochum-Langendreer - Universitätsklinik, Bochum
  - HELIOS Klinikum Erfurt, Erfurt
  - Universitätsklinikum Erlangen, Erlangen
  - Alfried Krupp Krankenhaus, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - LMU Klinikum der Universität München, Munich
  - Klinikum Nürnberg - Klinikum Nürnberg Süd, Nuremberg
- Hellenic Airforce 251 General Hospital, Athens, Greece
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - The University of Hong Kong, Hong Kong
- Országos Klinikai Idegtudományi Intézet, Budapest, Hungary
- Israel (2):
  - Hadassah Medical Organization, Jerusalem
  - Sheba Medical Center, Ramat Gan
- Italy (3):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedaliera Ospedale Niguarda Cà Granda, Milan
- Military Medical Institute-Wojskowy Instytut Medyczny, Warsaw, Poland
- Centro Hospitalar de Vila Nova de Gaia/Espinho - Unidade I, Vila Nova de Gaia, Portugal
- Russia (2):
  - Siberian Federal Biomedical Research Center, Novosibirsk
  - Almazov National Medical Research Centre, Saint Petersburg
- CINRE s.r.o., Bratislava, Slovakia
- Chris Hani Baragwaneth Hospital, Johannesburg, South Africa
- South Korea (9):
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - Jeonbuk National University Hospital, Jeonju
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Ajou University Medical Center, Suwon
  - Ulsan University Hospital, Ulsan
- Spain (9):
  - Hospital De Cruces, Barakaldo
  - Hospital Vall D'Hebron, Barcelona
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Álvaro Cunqueiro, Vigo
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - Inselspital - Universitätsspital Bern, Bern
  - Hôpitaux Universitaires de Genève, Geneva
- Cleveland Clinic - Abu Dhabi, Abu Dhabi, United Arab Emirates
- United Kingdom (5):
  - University Hospitals of Birmingham NHS Foundation Trust - Queen Elizabeth Hospital, Birmingham
  - Royal Infirmary of Edinburgh, Edinburgh
  - Imperial College Healthcare NHS Trust - Charing Cross Hospital, London
  - Barking, Havering and Redbridge University Hospitals - Queen's Hospital, Romford
  - University Hospitals of North Midlands NHS Trust - Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No
Only multi center data will be available